CLINICAL TRIAL: NCT01898754
Title: Drug-resistance Testing in Kenya to Improve ART Suppression of HIV Replication
Brief Title: Oligonucleotide Ligation Assay (OLA) Resistance Study
Acronym: OLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other); University of Nairobi (Other)
Responsible Party: Principal Investigator, Michael Chung, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14124-SCH
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: HIV Positive
Keywords: Transmitted Drug Resistance
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-ART Oligonucleotide Assay (OLA) (Experimental): Pre-ART OLA will be tested for resistance at 5 pol codons conferring high-level resistance to NNRTI and 3TC (K103N, V106M, Y181C, G190A and M184V)
  Interventions: Other: Pre-ART Oligonucleotide Assay (OLA)
- No OLA (Standard of Care [SOC]) (No Intervention): The participants will receive standard of care as per Kenya guidelines but will be offered OLA resistance testing after 12 months

INTERVENTIONS:
Other: Pre-ART Oligonucleotide Assay (OLA) — Block randomization (1:1) to pre-ART OLA testing or OLA testing after 12mo on ART
  Other Names: Pre-ART OLA
  Arms: Pre-ART Oligonucleotide Assay (OLA)

SUMMARY:
The investigators propose to gauge improvements in the rate of durable suppression of viral replication by ART when OLA is used to guide clinical decisions at the PEPFAR Coptic Hope Center in Kenya, and to determine the cost-effectiveness of implementing this strategy at Coptic Hope Center.

DETAILED DESCRIPTION:
Durable suppression of HIV replication is critical to (1) improving the health of infected individuals, (2) to reducing HIV transmission to sexual partners and from mothers to their infants, and (3) to maintaining the effectiveness of the current 1st-line non-nucleoside reverse transcriptase inhibitors (NNRTI)- based ART. Across multiple trials, individuals with NNRTI-resistance, even at low-concentrations, have substantially greater virologic failure when treated with NVP- vs PI-ART. A cost-effective strategy is needed to detect and manage ARV-resistant HIV infections. A simple low-cost innovative assay the investigators developed and successfully transferred to Asian and African countries (oligonucleotide ligation assay (OLA)) can detect NNRTI+lamivudine (3TC) resistant HIV using reagents that costs <$7.00/person. Furthermore, detection of NNRTI-resistance by OLA is highly (P<0.001) associated with virologic failure of nevirapine (NVP)-ART in two retrospective studies; one of Thai women who had been previously randomized to single-dose NVP and the second of ARV-naïve Kenyan adults.

The investigators hypothesize that implementation of OLA into routine care will allow Kenyan clinicians to appropriately target protease inhibitor (PI)-based ART and improve rates of durable suppression of viral replication, and thus improve CD4 cell gains and individuals' health, reduce the transmission of ARV-resistant HIV within the community, and maintain the utility of NNRTI-ART. In addition, the investigators hypothesize that programmatically OLA-guided ART will be more cost-efficient compared to the current strategy of empiric use of NNRTI-ART as initial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection
2. >2 years of age
3. Qualifying for 1st-line ART based on Kenyan Guidelines
4. Plan to reside in area for >1 year
5. Adult patient or parent of minor agrees to study and provides informed consent

Exclusion Criteria:

1. Received ART previously from Hope Center
2. Ongoing ART
3. Plan to start 2nd-line ART

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Frenkel, MD, Principal Investigator — University of Washington, Seattle Children's Research Institute; Michael H Chung, MD, MPH, Principal Investigator — Department of Global Health, University of Washington
Locations (2):
- Kenya (2):
  - Coptic Hospital, Maseno
  - Coptic Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung MH, McGrath CJ, Beck IA, Levine M, Milne RS, So I, Andersen N, Dross S, Coombs RW, Chohan B, Yatich N, Kiptinness C, Sakr SR, Kiarie JN, Frenkel LM. Evaluation of the management of pretreatment HIV drug resistance by oligonucleotide ligation assay: a randomised controlled trial. Lancet HIV. 2020 Feb;7(2):e104-e112. doi: 10.1016/S2352-3018(19)30337-6. Epub 2019 Dec 7. PMID 31818716
- [Derived] Silverman RA, Beck IA, Kiptinness C, Levine M, Milne R, McGrath CJ, Bii S, Richardson BA, John-Stewart G, Chohan B, Sakr SR, Kiarie JN, Frenkel LM, Chung MH. Prevalence of Pre-antiretroviral-Treatment Drug Resistance by Gender, Age, and Other Factors in HIV-Infected Individuals Initiating Therapy in Kenya, 2013-2014. J Infect Dis. 2017 Dec 19;216(12):1569-1578. doi: 10.1093/infdis/jix544. PMID 29040633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Started | 494 | 497
Received OLA or SOC as Randomly Assigned | 492 (2 participants did not receive OLA [1 died; 1 participant was HIV-uninfected]) | 495 (2 participants did not receive SOC [1 lost to follow-up prior to ART initiation; 1 participant was HIV-uninfected])
Completed | 400 | 403
Not Completed | 94 | 94

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC]) | Total
Number analyzed (Participants) | 492 | 495 | 987
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [32 to 46] | 37 [30 to 45] | 37 [31 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 320 | 321 | 641
  Male | 172 | 174 | 346
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 492 | 495 | 987
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 492 | 495 | 987

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Failure With OLA-guided ART vs. Standard of Care
Description: The primary endpoint will be a comparison of the rates of viral non-suppression >400 copies/mL between study arms at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 400 | 403
Participants | 34 | 39

2. Secondary Outcome: The Difference in Virologic Failure Among Participants With Transmitted Drug-resistance (TDR) ≥10% Associated With Use of OLA-guided ART vs. SOC
Description: We did not analyze and report outcome of people with TDR ≥10%, instead we reported pretreatment drug resistance (PDR) as this parameter could be determined but antiretroviral history was not reliably available. Thus, PDR ≥10% is considered below in place of TDR ≥10%.
  Chung et al. Lancet HIV 2020; 7: e104-12.
Time Frame: 15 months
Population: WHO defines pretreatment HIV drug resistance (PDR) as "DR that is detected in ARV drug-naive people initiating ART or people with prior ARV drug exposure initiating or reinitiating first-line ART. PDR is either transmitted or acquired drug resistance, or both". Thus, we did not report outcomes with TDR, instead we reported PDR as this could be determined but antiretroviral history was not available. Thus, PDR is reported in place of TDR. This included participants with PDR ≥10% at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 35 | 26
Participants
  Participants with PDR and virologic failure | 5 | 13
  Participants with PDR and no virologic failure | 30 | 13

3. Secondary Outcome: Difference in Virologic Failure in the Subgroup of Participants With Prior or Ongoing ART Use Associated With Use of OLA-guided ART vs. SOC
Description: The primary outcome was virologic failure defined as plasma HIV RNA of at least 400 copies per mL after initiation of antiretroviral therapy (ART).
Time Frame: 15 months
Population: The analysis population included only those participants that had prior or ongoing ART use (non-ARV naive) at randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-ART Oligonucleotide Assay (OLA) With Prior ART Use: Pre-ART OLA will be tested for resistance at 5 pol codons conferring high-level resistance to NNRTI and 3TC (K103N, V106M, Y181C, G190A and M184V). This analysis included those in the OLA arm with prior ART use.
- No OLA (Standard of Care [SOC]) With Prior ART Use: The participants will receive standard of care as per Kenya guidelines but will be offered OLA resistance testing after 12 months. Pre-This analysis included those in the SOC arm with prior ART use.
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) With Prior ART Use | No OLA (Standard of Care [SOC]) With Prior ART Use
Number analyzed (Participants) | 32 | 32
Participants
  Participants with pre-ART and virologic failure | 1 | 1
  Participants with pre-ART and no virologic failure | 31 | 31

4. Secondary Outcome: Prevalence of TDR by Consensus Sequencing and OLA
Description: We did not analyze and report outcome of people with TDR, instead we reported pretreatment drug resistance (PDR) as this parameter could be determined but antiretroviral history was not reliably available. Thus, PDR is considered below in place of TDR. PDR was assessed by OLA and confirmed by consensus sequence or next-generation sequencing.
Time Frame: 15 months
Population: WHO defines pretreatment HIV drug resistance (PDR) as "DR that is detected in ARV drug-naive people initiating ART or people with prior ARV drug exposure initiating or reinitiating first-line ART". Thus, we did not report outcomes with TDR, instead we reported PDR as this could be determined but antiretroviral history was not available. Thus, PDR is reported in place of TDR.
  This analysis included participants with PDR assessed by OLA and confirmed by consensus sequencing by study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 492 | 495
Participants
  Participants with PDR | 51 | 42
  Participants without PDR | 441 | 453

5. Secondary Outcome: Proportion of Subgroup With TDR With Virologic Failure by Randomization Arm
Description: We did not analyze and report outcome of people with TDR, instead we reported pretreatment drug resistance (PDR) as this parameter could be determined but antiretroviral history was not reliably available. Thus, PDR is considered below in place of TDR. The primary outcome for this analysis was the difference in virologic failure, defined as plasma HIV-1 RNA of at least 400 copies per mL following ART initiation, by PDR. [Chung et al. Lancet HIV 2020; 7: e104-12]
Time Frame: 15 months
Population: WHO defines pretreatment HIV drug resistance (PDR) as "DR that is detected in ARV drug-naive people initiating ART or people with prior ARV drug exposure initiating or reinitiating first-line ART". Thus, we did not report outcomes with TDR, instead we reported PDR as this could be determined but antiretroviral history was not available. Thus, PDR is reported in place of TDR.
  The population included the subgroup of participants with PDR in each study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 35 | 26
Participants
  Participants with PDR and virologic failure | 5 | 13
  Participants with PDR and no virologic failure | 30 | 13

6. Secondary Outcome: Estimates of Medical Resource Utilization During the One-year Trial Period
Description: Estimates of medical resource utilization during was not calculated. No data available (data on medical resource utilization was not collected during the one-year trial)
Time Frame: 15 months
Population: No data available (data on medical resource utilization was not collected).
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: An Assessment of the Potential Long-term Cost-effectiveness of OLA-guided Testing Over a Patient's Lifetime
Description: This was not calculated as the model could not test for a period longer than 15 years due to computing limitations.
Time Frame: 15 months
Population: This was not calculated as the model could not test for a period longer than 15 years due to computing limitations.
Groups:
- Costing Analysis: This was not calculated as the model could not test for a period longer than 15 years due to computing limitations.
Arm/Group | Costing Analysis
Number analyzed (Participants) | 0

8. Secondary Outcome: Determination of Whether Low-level ARV Resistance (<5%) Detected by PYRO But Not by OLA is Associated With Virologic Failure
Description: The prespecified outcomes of this study included differences in the rate of virologic failure over 24 months of efavirenz-based ART between participants by frequency of drug-resistant variants detected by next-generation sequencing at enrollment. Drug-resistance frequency was defined as the proportion of a nucleotide variant encoding a drug-resistant codon in specimens with at least 100 viral templates sequenced. Virologic failure was defined as plasma HIV RNA of at least 400 copies/ml in sequential specimens or at the final study visit in participants prescribed efavirenz-based ART. [Milne et al. AIDS 2022 Nov 15;36(14):1949-1958]
Time Frame: 24 months
Population: Analysis included 352 participants from Nairobi, including 332 with virologic suppression at month-12 of efavirenz-based ART who enrolled for a second year and 20 participants who experienced virologic failure by month-12 of efavirenz-based ART. Pretreatment drug-resistance was classified as: wild-type (0%), low-frequency (1-9%), high-frequency (10-100%). Virologic failure by month-24 of efavirenz-based ART, was compared between individuals with and without pretreatment drug-resistance.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Viral Suppression at 24 Months of ART; Participants With Virologic Failure by 24 Months of ART: Participants from the Nairobi Coptic Clinic included in 24-month follow up.
Arm/Group | Participants With Viral Suppression at 24 Months of ART | Participants With Virologic Failure by 24 Months of ART
Number analyzed (Participants) | 322 | 30
Participants
  Wild-type resistance | 301 | 20
  Low-frequency resistance | 10 | 5
  High-frequency resistance | 11 | 5

9. Other Pre Specified Outcome: Descriptions of Technology Transfer of OLA to the Hope Center Laboratory, Including Intra- and Inter-assay the Reproducibility, and Discussion of Obstacles and Possible Solutions
Description: Technology transfer of OLA to the Hope Center Laboratory in Kenya is described, including intra- and inter-assay the reproducibility, and discussion of obstacles and possible solutions.
  Duarte et a. AIDS 2018, 32:2301-2308
Time Frame: 15 months
Population: Technology transfer to Kenya is described, including quality control measures and a discussion of issues.
  Duarte et a. AIDS 2018, 32:2301-2308
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: A Comparison of OLA Results Obtained Using DBS in Kenya to Retesting of Same Specimens With Input of Viral Templates Measured in Seattle
Description: DBS were not tested in Kenya and thus, the comparison of OLA results obtained using DBS in Kenya to retesting of same specimens with input of viral templates measured in Seattle was not evaluated.
Time Frame: 15 months
Population: DBS were not tested in Kenya.
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Detection of Resistance Mutations at OLA Codons by OLA vs. Consensus Sequencing
Description: Rates of pre-treatment drug resistance among all study participants in the study were assessed by OLA but not by consensus sequencing (CS) due to the high cost of sequencing the entire population. However, all mutations detected by OLA were confirmed by CS in Seattle, and if not detected by CS were confirmed by next generation Illumina sequencing. Participants with any indeterminate OLA results were also sequenced to determine the genotype at the indeterminate codon.
Time Frame: Enrollment
Population: Among the subgroup of enrollment samples with both OLA and CS testing, we compared mutation detection by each method at OLA codons and assessed mutations at non-OLA codons detected by CS. Only mutations with Stanford HIVDR Program drug resistance mutation scores ≥10 were included.
Measure: Count of Participants; unit: Participants
Groups:
- Oligonucleotide Assay (OLA): Mutations detected by OLA at HIV reverse transcriptase codons 65, 103, 181, 184 and 190
- Consensus Sequencing (CS): Mutations detected by consensus sequencing in HIV reverse transcriptase
Arm/Group | Oligonucleotide Assay (OLA) | Consensus Sequencing (CS)
Number analyzed (Participants) | 475 | 475
Participants
  K103N | 69 | 44
  Y181C | 19 | 14
  G190A | 16 | 9
  K65R | 9 | 8
  M184V | 16 | 8
  Not detected | 346 | 392

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pre-ART Oligonucleotide Assay (OLA) | No OLA (Standard of Care [SOC])
All-Cause Mortality (participants affected / at risk) | 34/492 | 43/495
Serious Adverse Events (participants affected / at risk) | 39/492 | 34/495
Other Adverse Events (participants affected / at risk) | 32/492 | 26/495
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-ART Oligonucleotide Assay (OLA) (N=492) | No OLA (Standard of Care [SOC]) (N=495)
Anemia (Blood and lymphatic system disorders) | 3 | 4
Cryptococcal Meningitis (Infections and infestations) | 1 | 0
Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 4
Amoebiasis (Infections and infestations) | 1 | 0
Bell's Palsy (Nervous system disorders) | 0 | 1
Blocked Fallopian Tubes (Reproductive system and breast disorders) | 3 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Childbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 2
Esophageal Candidiasis (Infections and infestations) | 0 | 1
Fibroids (Reproductive system and breast disorders) | 1 | 0
Gastric Ulcers (Gastrointestinal disorders) | 1 | 0
Gastrointestinal distress (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hemorrhoidectomy (Gastrointestinal disorders) | 0 | 1
Hysterectomy (Reproductive system and breast disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Kaposi Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Low Blood Pressure (Cardiac disorders) | 0 | 1
Menigitis (Infections and infestations) | 1 | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Peptic Ulcer Disease (Gastrointestinal disorders) | 3 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rectal Bleeding (Gastrointestinal disorders) | 0 | 1
Road Traffic Accident (Musculoskeletal and connective tissue disorders) | 3 | 0
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tuberculosis (Infections and infestations) | 5 | 5
Threatened Abortion (Reproductive system and breast disorders) | 1 | 0
Thyroidectomy (Endocrine disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-ART Oligonucleotide Assay (OLA) (N=492) | No OLA (Standard of Care [SOC]) (N=495)
Bloating (Gastrointestinal disorders) | 1 | 0
Bloody Stool (Gastrointestinal disorders) | 0 | 1
Blurred Vision (Eye disorders) | 0 | 2
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Childbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Genital Ulcer (Infections and infestations) | 1 | 0
Goiter (Endocrine disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lip Swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Malaria (Infections and infestations) | 5 | 2
Mouth Ulcer (Gastrointestinal disorders) | 1 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1
Paresthesia (Nervous system disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Road Traffic Accident (Musculoskeletal and connective tissue disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tuberculosis (Infections and infestations) | 3 | 1
Tonsilitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No